CLINICAL TRIAL: NCT03740555
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single and Multiple Ascending Doses (SAD/MAD) Study Following Intravenous Administration in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of HNC042.
Brief Title: A Study of HNC042 in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNC042-101
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HNC042 single dose (Experimental): HNC042,freeze-dried powder,single ascending doses Single dose,
  Interventions: Drug: HNC042 single dose
- Placebo single dose (Placebo Comparator): Placebo single ascending doses , Intravenous route Single dose
  Interventions: Drug: Placebo single dose
- HNC042 multiple ascending doses (Experimental): HNC042,freeze-dried powder,multiple ascending doses, Intravenous route
  Interventions: Drug: HNC042 multiple ascending doses
- Placebo, multiple ascending doses (Placebo Comparator): Placebo, multiple ascending doses, Intravenous route,
  Interventions: Drug: Placebo multiple ascending doses

INTERVENTIONS:
Drug: HNC042 single dose — HNC042,freeze-dried powder,single ascending doses Single dose, Intravenous route,starting dose of 100mg escalating up to 1200mg
  Arms: HNC042 single dose
Drug: Placebo single dose — Placebo single ascending doses , Intravenous route Single dose, matching placebo
  Arms: Placebo single dose
Drug: HNC042 multiple ascending doses — HNC042,freeze-dried powder,multiple ascending doses, Intravenous route Multiple doses, daily for 7 days, anticipated doses: 300mg to 1200mg
  Arms: HNC042 multiple ascending doses
Drug: Placebo multiple ascending doses — Placebo, multiple ascending doses, Intravenous route, Multiple doses, daily for 7 days, matching placebo
  Arms: Placebo, multiple ascending doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety , tolerability and pharmacokinetics after single ascending of HNC042 given to healthy subjects, compared to placebo. Also, the safety , tolerability and pharmacokinetics of multiple ascending of HNC042 given to healthy subjects daily for 7 days compared to placebo , will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, age 18-56 years
* BMI between 18-34 kg/m2,and body weight not less than 50.0kg.

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Between screening and 7 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after a single and multiple intravenous dose in healthy subjects in terms of adverse events
Number of subjects with abnormal laboratory | Between screening and 7days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after single and multiple intravenous dose in healthy subjects in terms of abnormal laboratory
Number of subjects with abnormal electrocardiogram | Between screening and 7 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after a single and multiple intravenous dose in healthy subjects in terms of abnormal electrocardiogram
Number of subjects with abnormal physical examination | Between screening and 7 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after a single and multiple intravenous dose in healthy subjects in terms of abnormal physical examination
Number of subjects with abnormal vital signs | Between screening and 7 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after a single and multiple intravenous dose in healthy subjects in terms of abnormal vital signs

SECONDARY OUTCOMES:
The amount of HNC042 in plasma | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of HNC042 in plasma over time - pharmacokinetics (PK) - after a single and multiple intravenous dose in healthy subjects
The amount of HNC042 in urine | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of HNC042 in urine over time - pharmacokinetics (PK) - after a single and multiple intravenous dose in healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo B. DePetrillo, Baltimore, Maryland, United States